CLINICAL TRIAL: NCT07278856
Title: Ruxolitinib in Combination With Chemotherapy for Untreated Nodal T-Follicular Helper (TFH) Cell Lymphomas
Brief Title: Ruxolitinib in Combination With CHOP Chemotherapy for the Treatment of Untreated Nodal T-Follicular Helper Cell Lymphomas
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25404; NCI-2025-08060 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25404 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-11-28; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Follicular Helper T-Cell Lymphoma; Follicular Helper T-Cell Lymphoma, Angioimmunoblastic-Type; Follicular Helper T-Cell Lymphoma, Follicular-Type; Follicular Helper T-Cell Lymphoma, Not Otherwise Specified; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Peripheral T-Cell Lymphoma, Not Otherwise Specified
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Specimen Handling; Biopsy; Cyclophosphamide; Doxorubicin; Filgrastim; Granulocyte Colony-Stimulating Factor; Fluorodeoxyglucose F18; pegfilgrastim; pegylated granulocyte colony-stimulating factor; Prednisone; deltacortene; prednylidene; ruxolitinib; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib, CHOP) (Experimental): See Detailed Description
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography; Biological: Filgrastim; Other: Fludeoxyglucose F-18; Procedure: Multigated Acquisition Scan; Biological: Pegfilgrastim; Drug: Prednisone; Other: Questionnaire Administration; Drug: Ruxolitinib Phosphate; Drug: Vincristine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT and FDG-PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: FDG-Positron Emission Tomography — Undergo FDG-PET/CT
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Biological: Filgrastim — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Other: Fludeoxyglucose F-18 — Given FDG
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Pegfilgrastim — Given SC
  Other Names: Dulastin; Filgrastim SD-01; filgrastim-SD/01; Fulphila; Fylnetra; G-Lasta; HSP-130; Jinyouli; Neulasta; Neulastim; Neupopeg; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; Pegfilgrastim-apgf; Pegfilgrastim-bmez; Pegfilgrastim-cbqv; Pegfilgrastim-fpgk; Pegfilgrastim-jmdb; Pegfilgrastim-pbbk; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Stimufend; Tripegfilgrastim; Udenyca; Ziextenzo
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Other: Questionnaire Administration — Ancillary studies
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi; Jakavi
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This phase I trial tests the safety, side effects and best dose of ruxolitinib in combination with cyclophosphamide, doxorubicin, vincristine, prednisone (CHOP) chemotherapy and how well the combination works in treating patients with untreated nodal T-follicular helper (TFH) cell lymphoma. Ruxolitinib phosphate blocks a protein called janus kinase, which may help keep abnormal blood cells or cancer cells from growing. It may also lower the body's immune response. Ruxolitinib phosphate is a type of tyrosine kinase inhibitor. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's deoxyribonucleic acid (DNA) and may kill cancer cells. It may also lower the body's immune response. Doxorubicin damages the cell's DNA and may kill cancer cells. It also blocks a certain enzyme needed for cell division and DNA repair. Doxorubicin is a type of anthracycline antitumor antibiotic. Vincristine is in a class of medications called vinca alkaloids. It works by stopping cancer cells from growing and dividing and may kill them. Prednisone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Giving ruxolitinib in combination with CHOP chemotherapy may be safe, tolerable, and/or effective in treating patients with untreated nodal TFH cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the safety of ruxolitinib phosphate (ruxolitinib) in combination with CHOP chemotherapy in untreated nodal TFH cell lymphoma patients.

SECONDARY OBJECTIVES:

I. Determine the tolerability and preliminary clinical efficacy of Ia. Ruxolitinib in combination with CHOP chemotherapy in untreated nodal TFH cell lymphoma; Ib. Ruxolitinib monotherapy maintenance for nodal TFH cell lymphoma patients who achieve a response (partial response [PR] or complete response [CR]) with ruxolitinib + CHOP chemotherapy.

EXPLORATORY OBJECTIVES:

I. Describe preliminary survival outcomes. II. Describe the relative dose intensity of CHOP chemotherapy backbone.

OUTLINE:

PART A: Patients receive ruxolitinib orally (PO) twice daily (BID) on days 1-21, cyclophosphamide intravenously (IV), doxorubicin IV, vincristine IV, on day 1 and prednisone PO once daily (QD) on days 1-5 of each cycle. Patients also receive pegfilgrastim subcutaneously (SC) 24-72 hours after last dose of treatment, filgrastim SC starting 1 day after last dose of treatment until absolute neutrophil count (ANC) > 1000/uL. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve a PR or CR and are ineligible for or decline consolidative autologous stem cell transplantation (ASCT) proceed to Part B.

PART B: Patients receive ruxolitinib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. After the first year of monotherapy maintenance, patients who remain in continuous CR or PR (compared to baseline imaging before Part A) may optionally continue to receive ruxolitinib for an additional 12 cycles.

Additionally, patients undergo bone marrow biopsy and aspiration and multigated acquisition scan (MUGA) or echocardiography (ECHO) at screening, blood sample collection, fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/computed tomography (CT) and CT throughout the study.

After completion of study treatment, patients are followed up at 30 days then for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document
* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Be ≥ 18 years of age on day of signing informed consent
* Have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale (PS) at time of enrollment. Patients with a performance status of 2 on the ECOG scale due to lymphoma may be eligible with principal investigator (PI) approval
* Histologically confirmed nodal T-follicular helper (TFH) cell lymphomas. Nodal TFH cell lymphomas include encompasses three subtypes:

  * Angioimmunoblastic T-cell lymphoma (AITL)(World Health Organization [WHO]4R)/follicular helper T-cell lymphoma (TFH lymphoma), angioimmunoblastic type (ICC)/nodal TFH cell lymphoma, angioimmunoblastic-type (WHO5)
  * Nodal peripheral T-cell lymphoma (PTCL) with TFH phenotype (nodal PTCL, TFH)(WHO4R)/TFH lymphoma, NOS (ICC)/nodal TFH cell lymphoma, not otherwise specified (NOS) (WHO5)
  * Follicular T-cell lymphoma (FTCL)(WHO4R)/TFH lymphoma, follicular type (ICC)/ nodal TFH cell lymphoma, follicular-type (WHO5)
* Must be planned to receive full course (6 cycles) chemoimmunotherapy as per clinical standard of care for untreated nodal TFH cell lymphoma
* Have measurable disease, including at least 1 nodal site measuring 1.5 cm or 1 extranodal site measuring 1.0 cm in longest dimension on CT or FDG-PET or marrow-only disease (disease only found on bone marrow biopsy)
* Left ventricular ejection fraction (LVEF) ≥ 50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3
* Hemoglobin ≥ 8 g/dL
* Platelets ≥ 100,000/mm^3 (≥ 50,000/mm^3 in cases of marrow infiltration by lymphoma or hypersplenism per investigator assessment)
* Measured or calculated creatinine clearance ≥ 60 mL/min (glomerular filtration rate [GFR] can also be used in place of creatinine clearance [CrCl])

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin ≤ 2.0 x upper limit of normal (ULN)

  * (Patients with documented liver or pancreatic involvement with lymphoma may be enrolled if total bilirubin ≤ 3.0 x ULN. Patients with documented Gilbert disease may be enrolled if total bilirubin ≤ 5.0 x ULN) OR direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3.0 x ULN OR ≤ 5 x ULN for patients with liver involvement
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN

  * Note: unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants, or patient is shown to have an antiphospholipid antibody on workup
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN

  * Note: unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants, or patient is shown to have an antiphospholipid antibody on workup
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of ≤ 1% per year during the treatment period and for at least 4 months after the last dose of study treatment. Women must refrain from donating eggs during this same period. A woman is considered to be of childbearing potential if she is post-menarchal, has not reached a postmenopausal state (≤ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements. Examples of contraceptive methods with a failure rate of ≤ 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception
* For women of childbearing potential, a negative serum pregnancy test result during screening period. Women who are considered not to be of childbearing potential are not required to have a pregnancy test
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 4 months after the last treatment. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of preventing drug exposure. Male patients considering preservation of fertility should bank sperm before study treatment
* TO BE ASSESSED UPON COMPLETION OF PART A FOR CONSIDERATION FOR PART B ONLY: Completion of first-line multi-agent chemotherapy with ruxolitinib with CHOP
* TO BE ASSESSED UPON COMPLETION OF PART A FOR CONSIDERATION FOR PART B ONLY: Documentation of response (PR or CR) per Lugano criteria within the previous 3 months
* TO BE ASSESSED UPON COMPLETION OF PART A FOR CONSIDERATION FOR PART B ONLY: Ineligible for or decline consolidative autologous stem cell transplantation. Ineligibility is defined by:

  * Patient deemed ineligible for high-dose chemotherapy and ASCT based on physician's assessment
  * AND at least one of the following criteria:

    * Age ≥ 65 years or
    * Age ≥ 18 years and Hematopoietic Cell Transplantation-specific Comorbidity Index (HCT-CI) score ≥ 3
* TO BE ASSESSED UPON COMPLETION OF PART A FOR CONSIDERATION FOR PART B ONLY: Recovery to ≤ grade 1 or baseline for any toxicities due to prior treatments, with the exception of peripheral neuropathy (recovery to ≤ grade 2) or alopecia

Exclusion Criteria:

* Contraindication to any of the individual components of CHOP, or if receiving an additional 6 cycles of anthracycline would place patient over the anthracycline lifetime cumulative dose (450 mg/m^2)
* Prior systemic treatment or radiation for T-cell lymphoma except for patients who require lymphoma symptom control during screening may receive steroids in the following manner:

  * Up to 30 mg/day of prednisone or equivalent may be used for lymphoma symptom control during screening, including prior to finalization of staging (not included as part of pre-phase treatment). If glucocorticoid treatment is urgently required at higher doses for lymphoma symptom control prior to the start of study treatment, tumor assessments must be completed prior to initiation of > 30-100 mg/day of prednisone or equivalent. Prednisone > 30-100 mg/day or equivalent may be given for a maximum of 7 days as a pre-phase treatment. If patients exceed the allowed dosing of corticosteroids, patients may still be eligible for the study provided that baseline imaging is performed (or repeated) after completion of the course of higher dose of steroids. Allowed corticosteroid dosing resets from the point of imaging forward and patients who do not exceed the allowed corticosteroid dosing from the point of imaging until initiation of study treatment may enroll
* Prior organ transplantation
* Known history of cirrhosis
* Current grade > 1 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease
* History of other malignancy that could affect compliance with the protocol or interpretation of results except with permission of the principal investigator. The following are eligible without a specific waiver:

  * Patients with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix at any time prior to the study are eligible
  * Patients with any malignancy appropriately treated with curative intent and the malignancy has been in remission without treatment for ≥ 2 years prior to enrollment are eligible
  * Patients with low-grade, early-stage prostate cancer (Gleason score 6 or below, stage 1 or 2) with no requirement for therapy at any time prior to study are eligible
* Evidence of significant, uncontrolled, concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* History of thrombosis, such as stroke or pulmonary embolism/deep vein thrombosis, within the last 6 months
* Recent major surgery (within 4 weeks prior to the start of cycle 1), other than for diagnosis
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block, or evidence of prior myocardial infarction in the last 6 months
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) which requires systemic treatment. Patients may proceed with screening during treatment for infection, but systemic treatment must be completed by cycle 1 day 1

  * If a patient has signs/symptoms suggestive of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, the patient must have a negative molecular (e.g., polymerase chain reaction [PCR]) test or 2 negative antigen test results at least 24 hours apart. Patients who do not meet SARS-CoV-2 infection eligibility criteria must be screen-failed and may only be rescreened if the following have been met:
  * At least 10 days since first positive test result have passed in asymptomatic patients or at least 10 days since recovery, defined as resolution of fever without use of antipyretics and improvement in symptoms
* Current and/or history of active tuberculosis or latent tuberculosis
* Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HBsAg] serology):

  * Patients with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HBsAg) may be included if hepatitis B virus (HBV) DNA is undetectable at the time of screening. These patients must be willing to undergo monthly DNA testing and appropriate antiviral therapy as indicated by institutional standard
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing)

  * Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History of uncontrolled HIV

  * Patients with known diagnosis of HIV must have undetectable viral load and be on anti-retroviral therapy
* Known human T cell lymphotropic virus (HTLV) 1/2
* Untreated latent tuberculosis
* Patients with known active central nervous system lymphoma
* Pregnancy or lactation or intending to become pregnant during study
* Symptomatic inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug (ruxolitinib) and/or predispose the subject to an increased risk of gastrointestinal toxicity
* Use of medications or consumption of foods that are strong inducers or inhibitors of cytochrome P450 (CYP)3A must be discontinued at least 2 weeks prior to study intervention. Patients who (after enrollment) require use of a strong CYP3A4 inhibitor to treat a fungal/mold infection will require dose reductions
* Participants who are receiving other investigational agents
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04-27 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ruxolitinib when given in combination with cyclophosphamide, doxorubicin, vincristine, prednisone (CHOP) chemotherapy | Prior to cycle 2 day 1 (cycle length = 21 days)
  Will be defined as the highest dose of ruxolitinib tested in which fewer than 33% of patients experience a dose-limiting toxicity and at least 6 patients have been treated at that dose. The MTD will be the recommended phase 2 dose, provided that other safety considerations are acceptable.
Incidence of adverse events | Up to 30 days after last dose of treatment
  Will be evaluated using Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Rate of ruxolitinib discontinuation due to toxicity while receiving ruxolitinib with CHOP therapy (Part A) | Up to 5 years
Complete response (CR) rate (Part A) | Up to 5 years
  A simple binary proportion and corresponding 95% confidence interval will be used to estimate CR.
Overall response rate (Part A) | Up to 5 years
  A simple binary proportion and corresponding 95% confidence interval will be used to estimate overall response.
Patient-reported outcomes (Part A) | Up to 30 days after last dose of study treatment
  Will be measured by the Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Health and Functional Assessment of Chronic Illness Therapy (FACT)-Item GP5 scale. Will be reported descriptively.
Rate of ruxolitinib discontinuation due to toxicity while receiving ruxolitinib maintenance monotherapy following ruxolitinib with CHOP (Part B) | Up to 5 years
Rate of conversion from partial response to CR (Part B) | Up to 5 years
Patient-reported outcomes (Part B) PROMIS | Up to 30 days after last dose of study treatment
  Will be measured by the PROMIS Global Health. Will be reported descriptively.
Patient-reported outcomes (Part B) FACT-Item GP5 | Up to 30 days after last dose of study treatment
  Will be measured by the FACT-Item GP5 scale. Will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Poh, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States